CLINICAL TRIAL: NCT02405702
Title: Does the Selection of Patients Helps Healing the Infection After Change in One Step of a Knee Replacement?
Brief Title: Importance of Patient Selection for Treatment of Infected Total Knee Prosthesis
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 007-14
Record Dates: First submitted 2015-01-25; First posted 2015-04-01 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Knee Infection
Keywords: Infection; Knee; knee replacement
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: restrospective study

SUMMARY:
The infection of a total knee replacement often imposes changing implants. The change in two step is currently considered the gold standard. The change in one step is a much debated attitude: strictly contra-indicated for some professionals, but others agree to reserve these for favorable suspected cases selected. Several criteria have been proposed in the literature: age, condition, duration of infection, known bacterium responsible, not virulent and sensitive to antibiotics, no fistula, no significant bone destruction. But these criteria are poorly validated, standing over an experience of surgical teams rather than high-level scientific studies. Some authors have proposed to achieve change in one step systematically. The results of these cohorts on healing the infection does not seem very different from the changes in two steps. But it is most often single-center series, uncontrolled, with small numbers.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patient having surgery for the management of knee infection after change in one step of a knee replacement prothesis in the participating services between 2000 and 2010.

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years having surgery for the management of knee infection after change in one step of a knee replacement prothesis in the participating services between 2000 and 2010.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Recovery from the infection measured visually | for the duration of hospital stay, up to 1 year
  show that the selection process of patients used improve treatment outcomes of infection in total knee replacement

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, Principal Investigator — University Hospital, Strasbourg, France